CLINICAL TRIAL: NCT06311578
Title: Phase 1 Study of Intratumoral Administration of JNJ-87704916, an Oncolytic Virus, as Monotherapy and in Combination for Advanced Solid Tumors
Brief Title: A Study of JNJ-87704916, as Monotherapy and in Combination for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Enterprise Innovation Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 87704916LUC1001; 2023-506495-27-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants with advanced solid tumors will receive JNJ-87704916 alone and in combination with cetrelimab. Ascending dose levels will be sequentially tested.
  Interventions: Drug: JNJ-87704916; Drug: Cetrelimab
- Part 2: Dose Expansion (Experimental): Part 2 will consist of two cohorts: Cohort A and Cohort B. Participants in both Cohorts with metastatic non-small cell lung cancer (NSCLC) will receive JNJ-87704916 in combination with cetrelimab at the dose identified in Part 1.
  Interventions: Drug: JNJ-87704916; Drug: Cetrelimab

INTERVENTIONS:
Drug: JNJ-87704916 — JNJ-87704916 will be administered as an intratumoral injection.
Drug: Cetrelimab — Cetrelimab will be administered.
  Other Names: JNJ-63723283

SUMMARY:
The purpose of this study is to determine the safety, feasibility, recommended dose(s) and regimen(s) of JNJ-87704916 as monotherapy and in combination with cetrelimab.

ELIGIBILITY:
Inclusion Criteria:

* For Part 1: Individuals with a diagnosis of advanced or metastatic solid tumor exhausting all available standard of care therapy; Part 2: Individuals with histologically or cytologically confirmed metastatic or locally advanced NSCLC
* Have at least 1 injectable tumor
* Eastern cooperative oncology group (ECOG) performance status of grade 0 or 1
* A participant who can have children must have a negative pregnancy test before the first dose of study treatment and during the study
* Thyroid function laboratory values within normal range except for participants on thyroid hormone replacement therapy

Exclusion Criteria:

* Active disease involvement of the CNS (example, primary central nervous system tumors, metastases, leptomeningeal disease). Some exceptions are allowed
* Prior history of, or active, significant herpetic infections (example, herpetic keratitis or encephalitis) or active herpetic infections that require ongoing systemic anti-viral therapy
* Active infection or condition that requires treatment with systemic anti-infective agents (example, antibiotics, antifungals, or antivirals) within 7 days prior to the first dose of study treatment or chronic use of anti-infective agents
* History of solid organ or hematologic stem cell transplantation
* Known positive test result for human immunodeficiency virus (HIV) or other immunodeficiency syndrome
* History of allergy to protein-based therapies or history of any significant drug allergy (such as anaphylaxis, hepatotoxicity, or immune-mediated thrombocytopenia or anemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2028-11-08 (Estimated); Study Completion 2032-08-26 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose-Limiting Toxicity (DLT) | Up to 5 years
  The DLTs are specific adverse events with defined non-hematological toxicities or hematologic toxicities as per the study protocol.
Number of Participants with Adverse Events (AEs) by Severity | From first dose up to 100 days after last dose of study treatment (up to 5 years)
  An adverse event is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the treatment. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening, and Grade 5: death related to adverse event.

SECONDARY OUTCOMES:
Parts 1 and 2: Percentage of Participants With Objective Response (OR) | Up to 5 years
  OR is defined as the percentage of participants who have best response of Complete Response (CR) or Partial Response (PR) according to response evaluation criteria in solid tumors (RECIST) v1.1.
Parts 1 and 2: Percentage of Participants With Disease Control (DC) | Up to 5 years
  DC is defined as the percentage of participants who have achieved complete response, partial response, and stable disease for at least 2 consecutive assessments according to RECIST v1.1.
Parts 1 and 2: Duration of Response (DOR) | Up to 5 years
  DOR will be calculated among responders from the date of initial documentation of a response to the date of first documented evidence of relapse according to RECIST v1.1, or death due to any cause, whichever occurs first.
Part 2: Progression Free Survival (PFS) | From treatment initiation until disease progression or worsening or death due to any cause (up to 5 years)
  PFS is defined as the time from treatment initiation until disease progression or worsening or death due to any cause.
Part 2: Overall Survival (OS) | From treatment initiation until death due to any cause (up to 5 years)
  OS is defined as the time from treatment initiation until death due to any cause.
Parts 1 and 2: Number of JNJ-87704916 Genome Copies per Milliliter | Up to 5 years
  Viral genome copies of JNJ-87704916 collected from samples (that is, blood, urine, oral mucosa, injection sites, and dressings) will be determined by quantitative polymerase chain reaction (qPCR) assays.
Parts 1 and 2: Payload Concentrations of JNJ-87704916 | Up to 2 years
  Blood samples will be collected to characterize JNJ-87704916 payload concentrations in blood will be analyzed using immunoassay.
Parts 1 and 2: Number of Participants with JNJ-87704916 Antibodies | Up to 2 years
  Antibodies against JNJ-87704916 encoded payloads and against herpes simplex virus type-1 (HSV-1) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Enterprise Innovation Inc Clinical Trial, Study Director — Johnson & Johnson Enterprise Innovation Inc.
Locations (9):
- United States (4):
  - NYU Langone Health, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Toronto General Hospital, Toronto, Ontario, Canada
- Gustave Roussy, Villejuif, France
- Spain (3):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency